CLINICAL TRIAL: NCT01471639
Title: A Prospective, Open-label, Nonrandomized Efficacy and Safety Trial of Intranasal Ketorolac in Emergency Department Patients for the Treatment of Acute Pain
Brief Title: An Efficacy and Safety Trial of Intranasal Ketorolac in Emergency Department Patients for the Treatment of Acute Pain
Acronym: Sprix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUI-S4
Record Dates: First submitted 2011-11-04; First posted 2011-11-15 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Other Acute Pain
Keywords: 18 years and older,; previously healthy; men and nonpregnant women; emergency department
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Emergencies | interventions — Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intranasal ketorolac (Sprix) (Experimental): FDA approved drug used in single arm study
  Interventions: Drug: intranasal ketorolac

INTERVENTIONS:
Drug: intranasal ketorolac — 15 mg
  Other Names: Sprix

SUMMARY:
The purpose of this study is to determine the effectiveness, the safety, and the tolerability of intranasal ketorolac (Sprix) in relieving acute pain in adults ages 18-65 who come to the ED seeking care. Considering all ED visits, pain is the most common chief complaint. Giving intranasal ketorolac (Sprix) after stomach and dental surgeries has been shown to be safe and effective, but no studies have investigated the use of intranasal ketorolac (Sprix) for the treatment of acute pain in the ED.

Ketorolac (Sprix) has several advantages over other drugs commonly given for pain, including opioids. Ketorolac (Sprix) is non-addicting and has fewer side effects than opioids. The administration of ketorolac (Sprix) by other methods, such as IV, intramuscular shot, and oral pill form, has been shown to be safe and effective in treating acute pain.

This study is being done to find out if giving ketorolac (Sprix) as a single dose nasal spray will have the same benefit in decreasing patient's pain.

DETAILED DESCRIPTION:
Adults between the ages of 18-65 were being seen in the emergency department of a single large tertiary care hospital with acute pain (moderate to severe 4-10 NRS scale). Those who met inclusion criteria were approached. Informed written consent was obtained from all participants. The study was approved by local Institutional Review Board (IRB). Demographics (age, gender, ethnicity) were recorded. Baseline pain scores on NRS were obtained prior to administration of the drug. Pain scores (NRS) after administration of the drug (intranasal ketorolac) were recorded. All adverse events/side effects were recorded. Data was obtained for the time the individual patient was in the emergency department being treated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is being seen in the emergency department (ED) in acute pain from an acute illness or injury (such as a kidney stone or an acute musculoskeletal injury)
2. Age ≥ 18 years and < 65 years
3. Stable patient with stable vital signs, including not in shock (systolic BP >90), not in respiratory failure, and not a multiple trauma patient
4. Mentally competent patient is able to understand the consent form
5. Baseline pain score is moderate to severe (e.g. on NRS ≥ 4 on a 0 to 10 NRS or ≥ 40 on a 0 to 100 NRS)

Exclusion Criteria:

1. Unstable patients
2. Multiple trauma patients
3. Patients with any allergies to ketorolac or any of the components in the nasal spray preparation
4. Patients with active peptic ulcer disease
5. Patients with a history of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDS
6. Patients about to undergo major surgery
7. Patients with renal disease or at risk for renal failure due to volume depletion
8. Pregnant or nursing mothers
9. Patients with suspected or confirmed cerebrovascular bleeding, patients with hemorrhagic diathesis, and/or those at high-risk of bleeding
10. Patient with a nasal abnormality or illness that could affect the absorption of intranasal medication (such as: nasal discharge, rhinitis, acute upper respiratory infection, acute epistaxis, nasal polyp, nasal tumor)
11. Patient with any other contraindication to the use of Sprix, or in whom use of Sprix would not be consistent with the approved package insert
12. History of chronic pain
13. History of drug abuse
14. History of significant neurologic disorder (could include diseases such as diabetic neuropathy, Parkinson's disease, etc)
15. History of significant psychiatric disorder
16. History of being on medications that may affect neurotransmitters (such as certain neurologic or psychiatric medications)
17. No immediate post-op patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Mace, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfaffenrath V, Fenzl E, Bregman D, Farkkila M. Intranasal ketorolac tromethamine (SPRIX(R)) containing 6% of lidocaine (ROX-828) for acute treatment of migraine: safety and efficacy data from a phase II clinical trial. Cephalalgia. 2012 Jul;32(10):766-77. doi: 10.1177/0333102412451359. Epub 2012 Jun 18. PMID 22711895

RESULTS

PARTICIPANT FLOW:
Recruitment Details: December 01, 2011 Emergency Department
Pre-assignment Details: Chronic pain, critical illness
Period: Overall Study
Arm/Group | Intranasal Ketorolac (Sprix)
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intranasal Ketorolac (Sprix)
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Intranasal Ketorolac on Numeric Pain Scale
Description: Change in numeric rating scale after receiving intranasal ketorolac. 0 (no pain) - 10 (worst possible pain)
Time Frame: up to 4 hours
Population: Improvement in pain score rating among participants rating from baseline pain scores, 20 minutes, 40 minutes, 1 hour, 2 hour, 3 hour and 4 hour post dose. Pain scale ranging from 0 (no pain) - 10 (worst possible pain)
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Ketorolac (Sprix)
Number analyzed (Participants) | 37
Participants
  Baseline: Reported Pain Score of 10 | 10
  Baseline: Reported Pain Score of 9 | 2
  Baseline: Reported Pain Score of 8 | 12
  Baseline: Reported Pain Score of 7 | 5
  Baseline: Reported Pain Score of 6 | 5
  Baseline: Reported Pain Score of 5 | 1
  Baseline: Reported Pain Score of 4 | 2
  Baseline: REported Pain Score of 3 | 0
  Baseline: Reported Pain Score of 2 | 0
  Baseline: Reported Pain Score of 1 | 0
  Baseline: Reported Pain Score of 0 | 0
  Baseline: No Rating | 0
  20 minutes: Reported Pain Score of 10 | 3
  20 minutes: Reported Pain Score of 9 | 2
  20 minutes: Reported Pain Score of 8 | 3
  20 minutes: Reported Pain Score of 7 | 2
  20 minutes: Reported Pain Score of 6 | 2
  20 minutes: Reported Pain Score of 5 | 6
  20 minutes: Reported Pain Score of 4 | 3
  20 minutes: REported Pain Score of 3 | 4
  20 minutes: Reported Pain Score of 2 | 5
  20 minutes: Reported Pain Score of 1 | 3
  20 minutes: Reported Pain Score of 0 | 4
  20 minutes: No Rating | 0
  40 minutes: Reported Pain Score of 10 | 2
  40 minutes: Reported Pain Score of 9 | 3
  40 minutes: Reported Pain Score of 8 | 3
  40 minutes: Reported Pain Score of 7 | 1
  40 minutes: Reported Pain Score of 6 | 1
  40 minutes: Reported Pain Score of 5 | 3
  40 minutes: Reported Pain Score of 4 | 2
  40 minutes: REported Pain Score of 3 | 1
  40 minutes: Reported Pain Score of 2 | 4
  40 minutes: Reported Pain Score of 1 | 1
  40 minutes: Reported Pain Score of 0 | 6
  40 minutes: No Rating | 10
  1 hour: Reported Pain Score of 10 | 1
  1 hour: Reported Pain Score of 9 | 0
  1 hour: Reported Pain Score of 8 | 1
  1 hour: Reported Pain Score of 7 | 0
  1 hour: Reported Pain Score of 6 | 0
  1 hour: Reported Pain Score of 5 | 1
  1 hour: Reported Pain Score of 4 | 0
  1 hour: REported Pain Score of 3 | 1
  1 hour: Reported Pain Score of 2 | 1
  1 hour: Reported Pain Score of 1 | 0
  1 hour: Reported Pain Score of 0 | 3
  1 hour: No Rating | 29
  2 hoiurs: Reported Pain Score of 10 | 0
  2 hoiurs: Reported Pain Score of 9 | 0
  2 hoiurs: Reported Pain Score of 8 | 1
  2 hoiurs: Reported Pain Score of 7 | 0
  2 hoiurs: Reported Pain Score of 6 | 0
  2 hoiurs: Reported Pain Score of 5 | 0
  2 hoiurs: Reported Pain Score of 4 | 0
  2 hoiurs: REported Pain Score of 3 | 0
  2 hoiurs: Reported Pain Score of 2 | 0
  2 hoiurs: Reported Pain Score of 1 | 0
  2 hoiurs: Reported Pain Score of 0 | 0
  2 hoiurs: No Rating | 36
  3 hours: Reported Pain Score of 10 | 0
  3 hours: Reported Pain Score of 9 | 1
  3 hours: Reported Pain Score of 8 | 0
  3 hours: Reported Pain Score of 7 | 0
  3 hours: Reported Pain Score of 6 | 0
  3 hours: Reported Pain Score of 5 | 0
  3 hours: Reported Pain Score of 4 | 0
  3 hours: REported Pain Score of 3 | 0
  3 hours: Reported Pain Score of 2 | 0
  3 hours: Reported Pain Score of 1 | 0
  3 hours: Reported Pain Score of 0 | 0
  3 hours: No Rating | 36
  4 hours: Reported Pain Score of 10 | 0
  4 hours: Reported Pain Score of 9 | 0
  4 hours: Reported Pain Score of 8 | 0
  4 hours: Reported Pain Score of 7 | 0
  4 hours: Reported Pain Score of 6 | 0
  4 hours: Reported Pain Score of 5 | 0
  4 hours: Reported Pain Score of 4 | 0
  4 hours: REported Pain Score of 3 | 0
  4 hours: Reported Pain Score of 2 | 0
  4 hours: Reported Pain Score of 1 | 0
  4 hours: Reported Pain Score of 0 | 0
  4 hours: No Rating | 37

2. Secondary Outcome: Adverse Event/Side Effects
Description: Safety assessed by reporting of all adverse events and side effects.
Time Frame: Up to 4 hours
Population: Participants who reported discomfort or unpleasant feeling associated with use of intranasal ketorolac
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Ketorolac (Sprix)
Number analyzed (Participants) | 37
Participants
  Reported a "burning" feeling | 7
  No adverse event/Side effect reported | 30

ADVERSE EVENTS:
Time Frame: 7 months
Description: Definition same as Clinicaltrials.gov.
Arm/Group | Intranasal Ketorolac (Sprix)
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 7/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Ketorolac (Sprix) (N=37)
Discomfort (burning feeling of nasal mucosa) (Skin and subcutaneous tissue disorders) | 7 (7) — 7 individual felt discomfort (a burning feeling) of the nasal mucosa. This resolved quickly, within minutes. Inspection of the nasal mucosa showed no visible abnormalities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-09-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT01471639/Prot_SAP_000.pdf
  • Informed Consent Form (2011-09-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT01471639/ICF_001.pdf